CLINICAL TRIAL: NCT04597385
Title: A Long-term Follow-up Study to Evaluate the Safety and Efficacy of RGX-121
Brief Title: Long-term Follow-Up for RGX-121
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGX-121-5101
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Mucopolysaccharidosis II
Keywords: MPS II; Gene Therapy; Hunter
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long-term Follow-Up: No intervention.
  Interventions: Other: Long-term Follow-Up

INTERVENTIONS:
Other: Long-term Follow-Up — No intervention

SUMMARY:
RGX-121-5101 is the long-term follow-up study to the RGX-121-101 first in human study where participants received RGX-121, a gene therapy intended to deliver a functional copy of the iduronate-2-sulfatase gene (IDS) to the central nervous system. This study will evaluate the long-term safety and efficacy of RGX-121.

DETAILED DESCRIPTION:
This is a prospective follow-up study to evaluate the long-term safety and efficacy after a single administration of RGX-121. Eligible participants are those who previously have enrolled in clinical study RGX-121-101 and received a single intracisternal (IC) or intracerebroventricular (ICV) infusion of RGX-121. Enrollment of each participant will occur the same day or after the participant has completed the end of study (EOS) visit or early termination visit (ET) from the previous (parent) study. Participants will be followed in this study cumulatively for up to 5 years after RGX-121 administration (inclusive of the parent study) or until RGX-121 is commercially available in the participant's country, whichever occurs first. No treatment will be directed under this observational protocol. The total study duration for each participant may vary depending on when they enroll in the current study following RGX-121 administration in the parent study.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible, a participant must have previously received RGX-121 in a separate parent trial.
* Participant or participant's legal guardian(s) is/(are) willing and able to provide written, signed informed consent

Exclusion Criteria:

* Patient has not received RGX-121 previously in a separate parent trial.

Min Age: 28 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 12 subjects over the age of 28 months who have received RGX-121 in a previous study.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-03-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidences of Adverse Events over time. | 3 years
  Safety
Incidences of Serious Adverse Events over time | 3 year
  Safety

SECONDARY OUTCOMES:
Biomarkers [Time frame: 1 Month, 12 Months, 24 Months, 36 Months] | 3 years
  Change from baseline in Glycosaminoglycan levels (ng/mL)
Changes in neurodevelopmental parameters of cognitive function [Time Frame: 1 Month, 12 Months, 24 Months, 36 Months] | 3 years
  Change from baseline in neurodevelopment parameters of cognitive, behavioral and adaptive function as measured by the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III) or Kaufman Assessment Battery for Children, 2nd Edition (KABC-II).
Changes in neurodevelopmental parameters of cognitive function [Time Frame: 1 Month, 12 Months, 24 Months, 36 Months] | 3 years
  Change from baseline in neurodevelopment parameters of cognitive, behavioral and adaptive function as measured by the Mullen Scales of Early Learning (MSEL)
Changes in neurodevelopmental parameters of adaptive behavior function [Time Frame: 1 Month, 12 Months, 24 Months, 36 Months] | 3 years
  Vineland Adaptive Behavior Scales Second Edition (VABS-II)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Pittsburgh - UPMC: Program for Neurodevelopment in Rare Disorders, Pittsburgh, Pennsylvania, United States